CLINICAL TRIAL: NCT04626635
Title: A Phase 1/2 Study of REGN7075 (EGFRxCD28 Costimulatory Bispecific Antibody) in Combination With Cemiplimab in Patients With Advanced Solid Tumors
Brief Title: A Trial to Find Out How Safe REGN7075 is and How Well it Works in Combination With Cemiplimab for Adult Participants With Advanced Cancers
Acronym: COMBINE-EGFR-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R7075-ONC-2009; 2022-501234-37-00 (EU CTIS Number)
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: Variety of mixed advanced solid tumor types; First in Human (FIH)
MeSH Terms: interventions — cemiplimab; Bevacizumab; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Dose Escalation (Experimental): Variety of mixed advanced solid tumor types
  Interventions: Drug: REGN7075; Drug: Cemiplimab
- Dose Expansion A (Experimental): Triple Negative Breast Cancer (TNBC)
  Interventions: Drug: REGN7075; Drug: Cemiplimab
- Dose Expansion B (Experimental): Cutaneous Squamous Cell Carcinoma (CSCC)
  Interventions: Drug: REGN7075; Drug: Cemiplimab
- Dose Expansion C (Experimental): Non-Small Cell Lung Cancer (NSCLC)
  Interventions: Drug: REGN7075; Drug: Cemiplimab; Drug: Platinum-based doublet chemotherapy
- Dose Expansion D (Experimental): Head and Neck Squamous Cell Carcinoma (HNSCC)
  Interventions: Drug: REGN7075; Drug: Cemiplimab
- Dose Expansion E (Experimental): Microsatellite Stable-Colorectal Cancer (MSS-CRC), with Active Liver Metastases and/or Active Peritoneal Metastases
  Interventions: Drug: REGN7075; Drug: Cemiplimab
- Dose Expansion F (Experimental): MSS-CRC with Isolated Lung/Lymph Node Metastases (no active liver and no active peritoneal metastases)
  Interventions: Drug: REGN7075; Drug: Cemiplimab
- Dose Expansion G (Experimental): Epidermal Growth Factor Receptor (EGFR) -mutant NSCLC Post Third Generation tyrosine kinase inhibitor (TKI)
  Interventions: Drug: REGN7075; Drug: Cemiplimab; Drug: Platinum-based doublet chemotherapy
- Dose Expansion H (Experimental): EGFR-mutant NSCLC Post Third Generation TKI and Post Platinum-Doublet Chemotherapy
  Interventions: Drug: REGN7075; Drug: Cemiplimab
- Dose Expansion I (Experimental): Third-line (3L) MSS-CRC with Active Liver Metastases
  Interventions: Drug: REGN7075; Drug: Cemiplimab; Drug: Bevacizumab; Drug: Trifluridine-tipiracil
- Dose Expansion J (Experimental): 3L MSS-CRC without Active Liver Metastases
  Interventions: Drug: REGN7075; Drug: Cemiplimab; Drug: Bevacizumab; Drug: Trifluridine-tipiracil

INTERVENTIONS:
Drug: REGN7075 — Intravenous (IV) infusion or subcutaneous (SC) injection will be administered every week (QW) or every 3 weeks (Q3W)
  Other Names: marlotamig
Drug: Cemiplimab — Administered concomitantly Q3W by IV infusion or SC injection
  Other Names: REGN2810; Libtayo
Drug: Platinum-based doublet chemotherapy — Administered IV Q3W
  Arms: Dose Expansion C; Dose Expansion G
Drug: Bevacizumab — Administered per protocol
  Arms: Dose Expansion I; Dose Expansion J
Drug: Trifluridine-tipiracil — Administered per protocol
  Arms: Dose Expansion I; Dose Expansion J

SUMMARY:
This study is researching an investigational drug called marlotamig (REGN7075) by itself and in combination with cemiplimab with or without chemotherapy. The study is focused on patients with certain solid tumors that are in an advanced stage.

The aim of the study is to see how safe and tolerable marlotamig is by itself and in combination with cemiplimab (with or without chemotherapy), and to find out what is the best dose of marlotamig to be given to patients with advanced solid tumors when combined with cemiplimab (with or without chemotherapy). Another aim of the study is to see how effective marlotamig by itself, or in combination with cemiplimab (with or without chemotherapy), is at treating cancer patients.

The study is also looking at:

* Side effects that may be experienced by people taking marlotamig by itself and in combination with cemiplimab with or without chemotherapy
* How marlotamig works in the body by itself and in combination with cemiplimab with or without chemotherapy
* How much marlotamig is present in the blood when given by itself and in combination with cemiplimab with or without chemotherapy
* To see if marlotamig by itself and in combination with cemiplimab with or without chemotherapy works to treat cancer by controlling the proliferation of tumor cells to shrink the tumor
* Whether the body makes antibodies against the study drugs (marlotamig and cemiplimab) (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
2. Has histologically or cytologically confirmed cancer that meets criteria as defined in the protocol
3. Expansion Cohorts only: Is anti-Programmed cell Death protein-1 (PD-1)/Programmed cell Death Ligand-1 (PD-L1) naïve, defined as never having previously been treated with a drug that targets the PD-1
4. Has at least 1 lesion that meets study criteria as defined in the protocol
5. Willing to provide tumor tissue from newly obtained biopsy (at a minimum core biopsy) from a tumor site that has not been previously irradiated
6. Has adequate organ and bone marrow function as defined in the protocol
7. In the judgement of the investigator, has a life expectancy of at least 3 months

Key Exclusion Criteria:

1. Is currently participating in another study of a therapeutic agent
2. Has participated in any study of an investigational agent or an investigational device within 4 weeks of the first administration of study drug as defined in the protocol
3. Has received treatment with an approved systemic therapy within 4 weeks of the first administration of study drug or has not yet recovered (ie, grade 1 or baseline) from any acute toxicities
4. Has received recent anti-Epidermal Growth Factor Receptor (EGFR) antibody therapy as defined in the protocol
5. Has received radiation therapy or major surgery within 14 days of the first administration of study drug or has not recovered (ie, grade 1 or baseline) from adverse events
6. Has received any previous systemic, non-immunomodulatory biologic therapy within 4 weeks of first administration of study drug.
7. Has had prior anti-cancer immunotherapy within 5 half-lives prior to study drug as defined in the protocol
8. Has second malignancy that is progressing or requires active treatment as defined in the protocol
9. Has any condition requiring ongoing/continuous corticosteroid therapy (>10 mg prednisone/day or anti-inflammatory equivalent) within 1-2 weeks prior to the first dose of study drug as defined in the protocol
10. Has ongoing or recent (within 5 years) evidence of significant autoimmune disease or any other condition that required treatment with systemic immunosuppressive treatments as defined in the protocol
11. Has untreated or active primary brain tumor, Central Nervous System (CNS) metastases, leptomeningeal disease, or spinal cord compression
12. Has encephalitis, meningitis, organic brain disease (eg, Parkinson's disease) or uncontrolled seizures within 1 year prior to the first dose of study drug
13. Has any ongoing inflammatory skin disease as defined in the protocol

NOTE: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 933 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of Dose-Limiting Toxicities (DLTs) during the DLT period | Up to 6 weeks
  Dose escalation
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs) | Approximately 90 days from last dose; up to 5 years
  Dose escalation
Incidence and severity of Adverse Events of Special Interest (AESIs) | Approximately 90 days from last dose; up to 5 years
  Dose escalation
Incidence and severity of Serious Adverse Events (SAEs) | Approximately 90 days from last dose; up to 5 years
  Dose escalation
Incidence and severity of grade ≥3 laboratory abnormalities | Approximately 90 days from last dose; up to 5 years
  Dose escalation
Objective Response Rate (ORR) | Up to 5 years
  Dose expansion

SECONDARY OUTCOMES:
Concentrations of marlotamig in serum | Up to 5 years
  Dose escalation and dose expansion
ORR | Up to 5 years
  Dose escalation
Progression Free Survival (PFS) | Up to 5 years
  Dose escalation and dose expansion
Duration of Response (DOR) | Up to 5 years
  Dose escalation and dose expansion
Disease Control Rate (DCR) | Up to 5 years
  Dose escalation and dose expansion
Complete Response (CR) rate | Up to 5 years
  Dose escalation and dose expansion
Overall survival (OS) | Up to 5 years
  Dose escalation and dose expansion
Incidence of Anti-Drug Antibodies (ADA) to marlotamig | Approximately 90 days from last dose; up to 5 years
  Dose escalation and dose expansion
Magnitude of ADA to marlotamig | Approximately 90 days from last dose; up to 5 years
  Dose escalation and dose expansion
Incidence of ADA to cemiplimab | Approximately 90 days from last dose; up to 5 years
  Dose escalation and dose expansion
Magnitude of ADA to cemiplimab | Approximately 90 days from last dose; up to 5 years
  Dose escalation and dose expansion
The incidence and severity of TEAEs | Approximately 90 days from last dose; up to 5 years
  Dose expansion
The incidence and severity of AESIs | Approximately 90 days from last dose; up to 5 years
  Dose expansion
The incidence and severity of SAEs | Approximately 90 days from last dose; up to 5 years
  Dose expansion
The incidence and severity of grade ≥3 laboratory abnormalities | Approximately 90 days from last dose; up to 5 years
  Dose expansion
Patient reported Quality of Life (QoL) per European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 | Approximately 90 days from last dose; up to 5 years
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Patient reported Quality of Life (QoL) per EORTC QLQ-CR29 in CRC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ CR-29 questionnaire consists of 29 items (Likert scale), with a response scale for each of them from 1 to 4, with the following structure: 1 = Not at All 2 = A little; 3 = Quite a Bit; 4 = Very much. The QLQ-CR29 has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest (men), impotence, sexual interest (women), and dyspareunia). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Patient reported Quality of Life (QoL) per EORTC QLQ-BR23 in breast cancer patients | Approximately 90 days from last dose; up to 5 years
  The EORTC-QLQ-BR23 includes functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and single item symptoms scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). Questions use 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Scores average and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems.
Patient reported Quality of Life (QoL) per EORTC QLQ-LC13 in NSCLC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ-LC13 is a 13-item, disease-specific module which assesses quality of life across multiple scales, including dyspnea, cough and chest pain.
  The scale for EORTC-QLQ-LC13 is 1-4 for most outcome measures of systems, with 1 rated as "not at all" and 4 rated as "very much".
Patient reported Quality of Life (QoL) per EORTC QLQ-HN35 in HNSCC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ-HN35 is a 35-item, disease-specific module which assesses quality of life across multiple scales, including pain, swallowing, and senses.
  The questionnaire has 35 Likert type questions in total and the evaluation is made by giving the score of None: 1, A little: 2, Quite: 3, A lot: 4.
Patient reported Quality of Life (QoL) per EQ-5D-5L | Approximately 90 days from last dose; up to 5 years
  The EQ-5D-5L consists of EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Patient reported symptoms per EORTC QLQ-C30 | Approximately 90 days from last dose; up to 5 years
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Patient reported symptoms per EORTC QLQ-CR29 in CRC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ CR-29 questionnaire consists of 29 items (Likert scale), with a response scale for each of them from 1 to 4, with the following structure: 1 = Not at All 2 = A little; 3 = Quite a Bit; 4 = Very much. The QLQ-CR29 has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest (men), impotence, sexual interest (women), and dyspareunia). . Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Patient reported symptoms per EORTC QLQ-BR23 in breast cancer patients | Approximately 90 days from last dose; up to 5 years
  The EORTC-QLQ-BR23 includes functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and single item symptoms scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). Questions use 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Scores average and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems.
Patient reported symptoms per EORTC QLQ-LC13 in NSCLC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ-LC13 is a 13-item, disease-specific module which assesses quality of life across multiple scales, including dyspnea, cough and chest pain.
  The scale for EORTC-QLQ-LC13 is 1-4 for most outcome measures of systems, with 1 rated as "not at all" and 4 rated as "very much".
Patient reported symptoms per EORTC QLQ-HN35 in HNSCC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ-HN35 is a 35-item, disease-specific module which assesses quality of life across multiple scales, including pain, swallowing, and senses.
  The questionnaire has 35 Likert type questions in total and the evaluation is made by giving the score of None: 1, A little: 2, Quite: 3, A lot: 4.
Patient reported symptoms per EQ-5D-5L | Approximately 90 days from last dose; up to 5 years
  The EQ-5D-5L consists of EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Patient reported functioning per EORTC QLQ-C30 | Approximately 90 days from last dose; up to 5 years
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Patient reported functioning per EORTC QLQ-CR29 in CRC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ CR-29 questionnaire consists of 29 items (Likert scale), with a response scale for each of them from 1 to 4, with the following structure: 1 = Not at All 2 = A little; 3 = Quite a Bit; 4 = Very much. The QLQ-CR29 has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest (men), impotence, sexual interest (women), and dyspareunia). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Patient reported functioning per EORTC QLQ-BR23 in breast cancer patients | Approximately 90 days from last dose; up to 5 years
  The EORTC-QLQ-BR23 includes functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and single item symptoms scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). Questions use 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Scores average and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems.
Patient reported functioning per EORTC QLQ-LC13 in NSCLC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ-LC13 is a 13-item, disease-specific module which assesses quality of life across multiple scales, including dyspnea, cough and chest pain.
  The scale for EORTC-QLQ-LC13 is 1-4 for most outcome measures of systems, with 1 rated as "not at all" and 4 rated as "very much".
Patient reported functioning per EORTC QLQ-HN35 in HNSCC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ-HN35 is a 35-item, disease-specific module which assesses quality of life across multiple scales, including pain, swallowing, and senses.
  The questionnaire has 35 Likert type questions in total and the evaluation is made by giving the score of None: 1, A little: 2, Quite: 3, A lot: 4.
Patient reported functioning per EQ-5D-5L | Approximately 90 days from last dose; up to 5 years
  The EQ-5D-5L consists of EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Patient reporting general health status per EORTC QLQ-C30 | Approximately 90 days from last dose; up to 5 years
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Patient reporting general health status per EORTC QLQ-CR29 in CRC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ CR-29 questionnaire consists of 29 items (Likert scale), with a response scale for each of them from 1 to 4, with the following structure: 1 = Not at All 2 = A little; 3 = Quite a Bit; 4 = Very much. The QLQ-CR29 has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items (urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, anxiety, weight, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, sexual interest (men), impotence, sexual interest (women), and dyspareunia). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Patient reporting general health status per EORTC QLQ-BR23 in breast cancer patients | Approximately 90 days from last dose; up to 5 years
  The EORTC-QLQ-BR23 includes functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and single item symptoms scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). Questions use 4-point Likert scale (1 'Not at All' to 4 'Very Much'). Scores average and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems.
Patient reporting general health status per EORTC QLQ-LC13 in NSCLC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ-LC13 is a 13-item, disease-specific module which assesses quality of life across multiple scales, including dyspnea, cough and chest pain.
  The scale for EORTC-QLQ-LC13 is 1-4 for most outcome measures of systems, with 1 rated as "not at all" and 4 rated as "very much".
Patient reporting general health status per EORTC QLQ-HN35 in HNSCC patients | Approximately 90 days from last dose; up to 5 years
  The EORTC QLQ-HN35 is a 35-item, disease-specific module which assesses quality of life across multiple scales, including pain, swallowing, and senses.
  The questionnaire has 35 Likert type questions in total and the evaluation is made by giving the score of None: 1, A little: 2, Quite: 3, A lot: 4.
Patient reporting general health status per EQ-5D-5L | Approximately 90 days from last dose; up to 5 years
  The EQ-5D-5L consists of EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (55):
- United States (20):
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of California Los Angeles (UCLA) Medical Center, Los Angeles, California
  - The Regents of the University of California, San Francisco, San Francisco, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion - Lung Cancer Clinic, Aurora, Colorado
  - University of Florida Health, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dana Farber Cancer Institute Brookline Avenue, Boston, Massachusetts
  - START Midwest - Cancer & Hematology Centers of Western Michigan, PC, Grand Rapids, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute - 25th Ave, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Oncology And Hematology, San Antonio, Texas
  - University of Washington/Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (12):
  - Centre Leon Berard (CLB) - Centre de Recherche en Cancerologie Lyon-Est (CRCL), Lyon, Auvergne-Rhone
  - Centre Jean Perrin, Clermont-Ferrand, Auvergne-Rhône
  - Hopital Lyon Sud, Pierre-Bénite, Auvergne-Rhône
  - Centre Georges Francois Leclerc, Dijon, Bourgogne-Franche-Comté
  - Institut Claudius Regaud, IUCT-Oncopole, Toulouse, Haute-Garonne
  - Institut Bergonie, Bordeaux, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers, Nouvelle-Aquitaine
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - Centre Antoine Lacassagne, Nice, Provence Alpes Cote dAzur
  - Hospital Paris Saint-Joseph, Paris
  - Begin Army Instruction Hospital, Saint-Mandé, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region
- Israel (6):
  - Sheba Medical Center, Ramat Gan, Central District
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Erasmus MC, Rotterdam
- Poland (2):
  - Medpolonia Sp. z o.o., Poznan, Wielkopolska
  - Dom Lekarski SA, Szczecin, Zach
- Spain (8):
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Quiron Salud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Genesis Care Hospital San Francisco de Asis, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clinico Universitario - University of Valencia, Valencia
- Turkey (Türkiye) (5):
  - Baskent Universitesi, Yüreğir, Adana
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Istanbul University Cerrahpasa at Cerrahpasa Medical Faculty, Istanbul
  - Istanbul Medeniyet University - Prof Dr Suleyman Yalcin Sehir Hospital, Istanbul
  - Ciftlikkoy Campus Yenisehir Mersin, Mersin

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry),
  * the legal authority to share the data,
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/